CLINICAL TRIAL: NCT05259956
Title: The Impact of "3+1" Multidimensional Therapeutic Exercises on the Progression of Adolescent Idiopathic Scoliosis
Brief Title: Trial on Two Treatments for Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Aerospace Center Hospital (Other)
Responsible Party: Principal Investigator, Zhang Yafei, Principal Investigator, Peking University Aerospace Center Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP2022-50-507005
Record Dates: First submitted 2022-02-16; First posted 2022-03-02 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "3 plus 1" multidimensional exercise therapy (Experimental): The intervention consists of a Schroth-based exercise session and a manipulative therapy of pelvic asymmetry.
  Interventions: Behavioral: "3 plus 1" multidimensional exercise therapy
- Schroth based scoliosis specific exercise (Active Comparator): The intervention consists of the Schroth-based exercise session.
  Interventions: Behavioral: Schroth based scoliosis specific exercise

INTERVENTIONS:
Behavioral: Schroth based scoliosis specific exercise — The intervention is set to be delivered in a one-hour Schroth-based exercise session, with the frequency of twice a week for five weeks. The exercise consists of active auto-correction in 3D, stabilizing the corrected posture, and training in ADL.
  Arms: Schroth based scoliosis specific exercise
Behavioral: "3 plus 1" multidimensional exercise therapy — The intervention is set to be delivered in a 90-minute exercise session, with a frequency of twice a week for five weeks. The exercise consists of a one-hour Schroth-based exercise session and an additional 30-minute manipulative therapy of pelvic asymmetry.
  Arms: "3 plus 1" multidimensional exercise therapy

SUMMARY:
Adolescent Idiopathic scoliosis is a three-dimensional structural deformity of the spine and pelvic that occurs in children. More evidence has arisen to emphasize the important role played by pelvic asymmetry during the progression of scoliosis. The purpose of this study is to compare the effectiveness of pelvic adjustments accompanied with Schroth-based exercises, with the latter alone in adolescent idiopathic scoliosis, to assess the impact of pelvic asymmetry on the spinal three-dimensional parametric features in scoliosis.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis is the most common three-dimensional structural deformity of the spine among adolescence, the International Society on Scoliosis Orthopaedic and Rehabilitation Treatment recommend specific exercise therapy to delay the progression of scoliosis. Many specific exercise therapies are effective in reducing the angle of coronal scoliosis, but their efficiency in sagittal and axial deformities hasn't been convincing. Recent studies have found that the axial asymmetry of the pelvis may be involved in the pathogenesis of idiopathic scoliosis, but there is no clinical study on the treatment of scoliosis by correcting the axial torsion of the pelvis neither at home nor abroad. So in this study, "3 plus 1" multidimensional exercise therapy was applied to mild adolescent idiopathic scoliosis for the first time.

The present study is a single-center randomized controlled trial conducted at the department of rehabilitation medicine, Aerospace Center Hospital. The written Informed consent will be obtained from each patient and one of their parents before inclusion. Eligible subjects will be randomized by a 1:1 allocation ratio either to the experimental group, in which the "3 plus 1" multidimensional exercise therapy will be performed and pelvic correction technique was adopted to correct pelvic axial rotation, or the control group, in which they will receive the Schroth-based exercise therapy. Blinded assessments will be conducted at baseline and 6-month after the intervention, including the differences in three-dimensional structural parameters of pelvis and spine, such as the ratio of the iliac widths, SRS-22 questionnaire, etc, to compare the efficacy of two different groups in improving the three-dimensional balance of the spine and the quality of daily life in adolescent idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of adolescent idiopathic scoliosis; Age from 10 to 18 years; A Cobb angle of 10 to 25 degrees; All maturity levels (Risser sign of 0-5).

Exclusion Criteria:

* Non-idiopathic scoliosis, which is caused by a neuromuscular, neurological, congenital malformation, or trauma-related comorbidity; Having mental problems or other contraindications to exercise; Previous fractures, rheumatic diseases, or operation history of lower extremities; Previous or current brace or surgical treatments for scoliosis.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Ratio of Iliac Widths at 24th week | baseline and at 24th week
  Rotation in the transverse plane of pelvic seen on a spinal standing full-length posteroanterior radiograph.

SECONDARY OUTCOMES:
Change in Cobb Angle | baseline and at 24th week
  The largest coronal convex curve is measured by the Cobb method on a spinal standing full-length posteroanterior radiograph.
Change in Apical Vertebral Translation in Main Curves | baseline and at 24th week
  When an apical vertebra or disc is identified as the apex of the curve, the center of the vertebra or disc is identified by drawing a horizontal line through the vertebra or disc, apical translation of the disc is measured from the disc centroid to the center sacral vertical line (CSVL).
Change in Coronal Pelvic Tilt | baseline and at 24th week
  The vertical distance between the horizontal tangents of the highest point of the bilateral iliac crest.
Change in Apical Vertebral Rotation in Main curves | baseline and at 24th week
  The Nash and Moe method is used to determine vertebral rotation. The apical vertebral body is divided into six equal segments longitudinally. When both pedicles are in view, there is no vertebral rotation. It is graded as "0". When the pedicle in the concave side (the right side) starts disappearing, it is graded as "1". When the pedicle disappears, it is graded as "2". When the contralateral pedicle (pedicle in the convex side) is in the midline of the vertebra, it is graded as "3". When it crosses the midline of the vertebra, it is graded as "4".
Change in Angle of Trunk Rotation | baseline and at 24th week
  The angle of trunk rotation will be measured with a Scoliometer.
Change in Scoliosis Research Society-22 Questionnaire | baseline and at 24th week
  The SRS-22 contains 22 questions covering 5 domains: function/activity 5 items; pain 5 items; self-perceived image 5 items; mental health 5 items; and satisfaction with treatment 2 items. Each item is scored from 1 (worst) to 5 (best). The sum of the 5 domains is 110.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Meng, Study Director — Aerospace Centre Hospital
Locations (1):
- Zhang yafei, Beijing, China